CLINICAL TRIAL: NCT01585376
Title: Study Recurrency Testing of Mutations Identified in WGS of Pediatric Rhabdomyosarcoma
Brief Title: Studying Genes in Samples From Younger Patients With Rhabdomyosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST12B3; COG-ARST12B3 (Other: Children's Oncology Group); ARST12B3 (Other: Children's Oncology Group); CDR0000732173 (Other: Clinical Trials.gov); NCI-2012-00729 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Sarcoma
Keywords: alveolar childhood rhabdomyosarcoma; embryonal childhood rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: mutation analysis
Genetic: nucleic acid sequencing
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and find biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

PURPOSE: This research trial studies genes in samples from younger patients with rhabdomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To obtain a larger cohort of rhabdomyosarcoma samples (alveolar and embryonal) to establish a more accurate estimate of the frequency of particular genetic lesions.
* To provide the statistical power to establish an unambiguous connection between focal genetic lesions, histological subtype, and outcome for patients with rhabdomyosarcoma.

OUTLINE: DNA samples are analyzed in solid and liquid phase for exons of all genes mutated from previous discovery. DNA is then eluted and sequenced by illumina platform.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Matched genomic deoxyribonucleic acid (DNA) from tumor and germline samples from patients diagnosed with rhabdomyosarcoma (alveolar or embryonal)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with rhabdomyosarcoma
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Frequency of particular genetic lesions
Identification of mutations that occur in at least 5% of rhabdomyosarcomas as a whole

CONTACTS AND LOCATIONS:
Overall Officials: Alberto S. Pappo, MD, Principal Investigator — St. Jude Children's Research Hospital